CLINICAL TRIAL: NCT05271981
Title: Uterine Artery Embolization For Uterine Pathology: What Impact On Fertility?
Brief Title: Fertility After Uterine Artery Embolization
Acronym: FERTI-EMBOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Gedeon Richter France (Unknown); Collège National des Gynécologues et Obstétriciens Français (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP21114; 2021-A01868-33 (Registry Identifier: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Fertility Disorders; Fertility Issues; Myoma;Uterus; Uterine Artery Embolisation
Keywords: uterine artery embolisation; Fertility Issues; Fertility Disorders; uterine myoma
MeSH Terms: conditions — Infertility; Myofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female who underwent uterine artery embolisation for uterine pathology
  Interventions: Other: Retrospective data collection; Other: Phone interview

INTERVENTIONS:
Other: Retrospective data collection — Data collection from the medical file of the patients
Other: Phone interview — Call for collecting fertility data and obstetrical issues of the patients

SUMMARY:
Uterine leiomyomas (or fibroids) are a common disease (30% of women over 35 years of age) in women of childbearing age and can cause various symptoms such as menometrorrhagia, dysmenorrhoea, pelvic pain and heaviness, and infertility.

Uterine artery embolisation, first used in France in 1990, is a safe, effective and less invasive therapeutic technique than surgical treatment (myomectomy or hysterectomy), particularly in the case of numerous and large fibroids. This technique is validated by the French National College of Gynaecologists-Obstetricians (CNGOF) as an alternative treatment for women who do not wish to become pregnant (grade A recommendation), but at present there is little reliable data concerning fertility, the occurrence of pregnancy and the obstetrical prognosis after uterine artery embolisation for fibroids. A recent systematic review of the literature with meta-analysis published very recently showed that 40.5% of patients with a desire for pregnancy were able to become pregnant after embolisation (CI: 33.3%-48.2%) but that the rates of miscarriage, obstetric complications and low birth weight were not negligible (respectively 33.5% (95% CI: 26.3-41%), 25.4% (95% CI = 13-40.2%) and 10% (95% CI = 6.2-14.6%) (Ghanaati et al. 2020).

In France, uterine artery embolisation is performed in more than thirty centres in women who have completed their parental project. On the other hand, in the absence of consistent literature, it is performed in patients of childbearing age, when it represents the only acceptable alternative or in the event of contraindication or refusal of surgery by the patient. To our knowledge, there is no large-scale French study to date on the impact of embolisation on fertility and pregnancy outcomes.

The aim of this study is to compile a retrospective database of all cases of uterine artery embolisation for uterine pathology performed at the Georges-Pompidou European Hospital (HEGP) since 2007 and to assess the impact of embolisation on fertility in patients of childbearing age.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years, ≤ 45 years at the time of their embolisation
* Uterine pathology responsible for disabling symptoms: uterine leiomyomas with no limitations in size, number or location, adenomyosis
* Having had a uterine artery embolisation between 2007 and September 2020
* Minimum delay of one year after embolisation
* Information and no opposition from patients

Exclusion Criteria:

* Women < 18 years and > 45 years at the time of embolisation
* Uterine artery embolisation for delivery haemorrhage
* Patients under court protection, guardianship or curatorship
* Refusal to participate in this research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female aged 18 to 45 years who underwent uterine artery embolisation for uterine pathology in our institution between 2007 and September 2020
Sampling Method: Probability Sample
Enrollment: 833 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Rate of live births after embolisation | one year
  Rate of live births after embolisation (percentage)

SECONDARY OUTCOMES:
Obstetrical outcomes after embolisation | one year
  * Pregnancy rate (percentage) ;
  * Miscarriage rate (percentage) ;
  * Assisted reproduction rate;
  * Obstetric complication rates (haemorrhage, caesarean section, prematurity, pre-eclampsia, placental disorders)
Effectiveness and safety of embolisation | one year
  * Complication rate of embolisation (percentage)
  * Post-embolisation myomectomy and hysterectomy rates (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Henri Azaïs, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlies results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Derived] Fabre C, Boeken T, Simon V, Dean C, Sapoval M, Pellerin O, Bats AS, Azais H, Koual M. Fertility outcomes after uterine artery embolization for symptomatic leiomyomas. CVIR Endovasc. 2025 Oct 16;8(1):83. doi: 10.1186/s42155-025-00604-4. PMID 41094296